CLINICAL TRIAL: NCT04823637
Title: Evaluating for a Correlation Between Osteopathic Examination and Ultrasonography on Thoracic Spine Asymmetry
Acronym: USOMM
Status: Completed | Type: Observational
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Randall Nydam, PhD, Associate Dean, Midwestern University
Other Study IDs: AZ 1232
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Osteopathic Manipulative Treatment; Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography vs Osteopathic manipulative medicine structural exam — Structural examination of the thoracic spine using ultrasound and osteopathic palpatory examination on skin.

SUMMARY:
Context: Thoracic spine is a common area of focus in osteopathic manipulative medicine (OMM) for a variety of conditions. Thoracic spine somatic dysfunction diagnosis is achieved by palpating for asymmetry at the tips of the transverse processes. Previous studies reveal that, instead of following the rule of threes, the transverse processes of a given thoracic vertebra generally align with the spinous process of the vertebra above. Ultrasonography has been widely used as a diagnostic tool to monitor musculoskeletal conditions. Ultrasound has the advantage of absence of radiation, and has shown comparable results to gold standard modalities like MRI in some areas of the spine. In the case of thoracic somatic dysfunction, ultrasound can be used to determine the location of each vertebral transverse process and its relationship with the spinous process. Previous studies have investigated the correlation between osteopathic manipulative medicine and ultrasonography of the cervical, lumbar, and sacral regions. However, no study has yet compared osteopathic structural examination with ultrasonographic examination of the thoracic vertebral region.

Objective: To determine whether there is a dependable correlation of osteopathic palpatory findings of the thoracic transverse processes with the measurements of ultrasonography.

Methods: Subjects were student volunteers recruited from the Midwestern University - Glendale campus. A non-toxic, non-permanent marker was used to mark bony landmarks on the skin to be used by the osteopathic examiners. Two osteopathic physicians (OMM1, OMM2) separately performed structural exams by palpating T2-T5 transverse processes to determine vertebral rotation. Two trained sonographers (US1, US2) separately scanned and measured the distance from the tip of the spinous process to the adjacent transverse processes of the vertebral segment below. Demographic variables were summarized with mean and standard deviation. Interexaminer reliability was assessed with percent agreement, Cohen's Kappa, and Fleiss' Kappa. Recruitment and protocols were approved by the MWU Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* First- and Second-year osteopathic medical students who received an email notification
* Masters program students who received an email notification

Exclusion Criteria:

- A history of or currently diagnosed with scoliosis, spondylosis, spondylolisthesis, herniated disc, spinal fracture, or surgery to the spine

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are Midwestern University students who were recruited via email announcements, with responses recorded via secure Google Form that was accessible only to the Midwestern University network.
  The overall demographics of participants showed 31 (47.0%) males and 35 (53.0%) females. Race and ethnicity were not collected for the purpose of this study as it was not a variable being evaluated or investigated. The subjects' age range is 22-35 years of age, with the mean age as 26.61 (SD = 3.1) for males and 25.71 (SD = 2.7) for females. The BMI range is 15.9 - 36.9kg/m2, with the mean BMI as 24.13 (SD = 4.2) overall, 25.46 (SD = 3.5) for males and 22.95 (SD = 4.5) for females.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Interexaminer reliability | Through study completion, which was an average of about 1 year
  We looked at the interexaminer reliability between ultrasound and osteopathic structural exam of the thoracic spine.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Nydam, PhD, Principal Investigator — Midwestern University
Locations (1):
- Midwestern University, Glendale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang S, Maddox J, Berg E, Kim K, Messier S, Swanson L, Dobrusin R, Stein AB, Nakken GN, Noble J, Nydam R. Evaluating for a correlation between osteopathic examination and ultrasonography on thoracic spine asymmetry. J Osteopath Med. 2021 Oct 13;122(1):31-43. doi: 10.1515/jom-2021-0020. PMID 34643344